CLINICAL TRIAL: NCT01959230
Title: A Single-Center, Double-Masked, Randomized, Vehicle-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Brimonidine Tartrate Ophthalmic Solution 0.025% Used Four Times Daily in a Population of Adult and Geriatric Subjects With Ocular Redness
Brief Title: Efficacy and Safety of Brimonidine Tartrate Ophthalmic Solution in Adult and Geriatric Participants With Ocular Redness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 861
Record Dates: First submitted 2013-10-08; First posted 2013-10-09 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Hyperemia
Keywords: Ocular redness
MeSH Terms: conditions — Hyperemia | interventions — Brimonidine Tartrate; Fluorescein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brimonidine Tartrate (Experimental): Participants will apply 1 drop of brimonidine tartrate ophthalmic solution 0.025% into each eye 4 times daily for up to 4 consecutive weeks.
  Interventions: Drug: Brimonidine Tartrate; Drug: Sodium Fluorescein; Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP
- Brimonidine Tartrate Vehicle (Placebo Comparator): Participants will apply 1 drop of the vehicle of brimonidine tartrate ophthalmic solution into each eye 4 times daily for up to 4 consecutive weeks.
  Interventions: Drug: Vehicle; Drug: Sodium Fluorescein; Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP

INTERVENTIONS:
Drug: Brimonidine Tartrate — Ophthalmic solution to be applied as directed.
  Arms: Brimonidine Tartrate
Drug: Vehicle — Ophthalmic solution to be applied as directed.
  Arms: Brimonidine Tartrate Vehicle
Drug: Sodium Fluorescein — For use as needed during the study for evaluating corneal damage.
Drug: Fluorescein Sodium and Benoximate Hydrocholoride Ophthalmic Solution USP — For use as needed during the study for intraocular pressure and dilated ophthalmoscopy.

SUMMARY:
To compare the efficacy and safety of brimonidine tartrate ophthalmic solution 0.025% with its vehicle for the treatment of ocular redness in a population of adult and geriatric participants with ocular redness.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Have a history of redness relief drops use or expressed a desire to use drops for redness relief, within the last 6 months.
* Have ocular health within normal limits including a calculated best-corrected visual acuity of 0.3 logarithm of the minimum angle of resolution (logMAR) or better in each eye, as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart.

Exclusion Criteria:

* Any ocular/systemic health problems.
* Use of any disallowed medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2013-12-20 (Actual); Study Completion 2013-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heleen DeCory, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Memphis, Tennessee, United States

REFERENCES:
- [Derived] McLaurin E, Cavet ME, Gomes PJ, Ciolino JB. Brimonidine Ophthalmic Solution 0.025% for Reduction of Ocular Redness: A Randomized Clinical Trial. Optom Vis Sci. 2018 Mar;95(3):264-271. doi: 10.1097/OPX.0000000000001182. PMID 29461408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive brimonidine tartrate ophthalmic solution or the vehicle of brimonidine tartrate ophthalmic solution, respectively.
Groups:
- Brimonidine Tartrate: Participants applied 1 drop of brimonidine tartrate ophthalmic solution 0.025% into each eye 4 times daily for up to 4 consecutive weeks.
- Brimonidine Tartrate Vehicle: Participants applied 1 drop of the vehicle of brimonidine tartrate ophthalmic solution into each eye 4 times daily for up to 4 consecutive weeks.
Period: Overall Study
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Started | 40 | 20
Received at Least 1 Dose of Study Drug | 40 | 20
Completed | 36 | 19
Not Completed | 4 | 1
Not completed — Failure to follow study procedures | 0 | 1
Not completed — Administrative reasons | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug (Safety Population).
Groups:
- Total: Total of all reporting groups
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (15.37) | 47.4 (15.36) | 47.5 (15.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 38
  Male | 18 | 4 | 22

OUTCOME MEASURES:

1. Primary Outcome: Ocular Redness as Measured by the Investigator Using the Ora Calibra™ Ocular Hyperemia Scale
Description: Ocular redness using the Ora Calibra Ocular Hyperemia Scale was scored by the Investigator using the following scale (allowing half unit increments): 0=None; 1.0=Mild-Slightly dilated blood vessels, color of vessels is typically pink, can be quadrantal; 2.0=Moderate-More apparent dilation of blood vessels, vessel color is more intense (redder), involves the majority of the vessel bed; 3.0=Severe-Numerous and obvious dilated blood vessels, in the absence of chemosis the color is deep red, may be less red or pink in presence of chemosis, is not quadrantic; 4.0=Extremely Severe-Large, numerous, dilated blood vessels characterized by unusually severe deep red color, regardless of grade of chemosis, which involves the entire vessel bed. A lower score is indicative of less redness.
Time Frame: 0 (predose), 5, 15, 30, 60, 90, 120, 180, and 240 minutes postdose on Day 1
Population: All randomized participants who received at least 1 dose of study drug and completed at least 1 post instillation ocular redness evaluation at Baseline (Intent-to-Treat [ITT] Population). Last Observation Carried Forward (LOCF) was used to impute missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 40 | 20
units on a scale
  Predose | 1.82 (0.412) | 1.71 (0.365)
  5 minutes Postdose | 0.58 (0.497) | 1.40 (0.666)
  15 minutes Postdose | 0.58 (0.497) | 1.35 (0.651)
  30 minutes Postdose | 0.59 (0.511) | 1.40 (0.641)
  60 minutes Postdose | 0.61 (0.509) | 1.40 (0.646)
  90 minutes Postdose | 0.60 (0.476) | 1.45 (0.672)
  120 minutes Postdose | 0.63 (0.470) | 1.53 (0.612)
  180 minutes Postdose | 0.73 (0.449) | 1.54 (0.586)
  240 minutes Postdose | 0.82 (0.474) | 1.54 (0.575)

2. Secondary Outcome: Ocular Redness as Measured by the Participant
Description: Ocular redness was scored daily pre-dose and post-dose on Days 1 to 29 and scored daily on Days 30 to 36 by the participant using a 0 to 4 unit scale (not allowing half unit increments). A lower score was indicative of less redness. The LOCF method used for this Secondary Outcome Measure was for imputing missing daily post-dose mean scores for entire days. If ≥1 score was provided for a day, imputation was not done. Imputation was done within the dosing period and separately within the follow-up period. The average (mean) daily pre-dose and post-dose scores for the dosing period Day 1 to Day 15 and dosing period Day 15 to Day 29, and the average (mean) daily score for the follow-up period Day 29 to Day 36 are reported.
Time Frame: Day 1 to Day 15; Day 15 to Day 29; Day 29 to Day 36
Population: All randomized participants who received at least 1 dose of study drug and completed at least 1 post instillation ocular redness evaluation at Baseline (ITT Population) with evaluable participant-recorded ocular redness data. LOCF method used as described in the Outcome Measure Description.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 40 | 20
units on a scale
  Daily Predose Score of Day 1 to Day 15: number analyzed (Participants) | 39 | 20
  Daily Predose Score of Day 1 to Day 15 | 1.52 (0.857) | 1.83 (0.975)
  Daily Postdose Score of Day 1 to Day 15: number analyzed (Participants) | 39 | 20
  Daily Postdose Score of Day 1 to Day 15 | 0.85 (0.860) | 1.85 (0.843)
  Daily Predose Score of Day 15 to Day 29: number analyzed (Participants) | 38 | 19
  Daily Predose Score of Day 15 to Day 29 | 1.45 (0.811) | 1.59 (1.012)
  Daily Postdose Score of Day 15 to Day 29: number analyzed (Participants) | 39 | 19
  Daily Postdose Score of Day 15 to Day 29 | 0.80 (0.810) | 1.63 (0.887)
  Daily Score of Day 29 to Day 36: number analyzed (Participants) | 36 | 19
  Daily Score of Day 29 to Day 36 | 1.69 (0.885) | 1.69 (0.897)

3. Secondary Outcome: Change From Predose Ocular Redness Score as Measured by the Investigator Using the Ora Calibra Ocular Hyperemia Scale
Description: as for outcome 1
Time Frame: 0 (predose), 1, 360, and 480 minutes (min) postdose on Day 1 and 0 (predose), 1, and 5 min postdose on Days 15 and 29
Population: All randomized participants who received at least 1 dose of study drug and completed at least 1 post instillation ocular redness evaluation at Baseline (ITT Population) with evaluable Investigator-recorded ocular redness data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Number analyzed (Participants) | 40 | 20
units on a scale
  Predose on Day 1 | 1.82 (0.412) | 1.71 (0.365)
  Change from Predose at 1 min Postdose on Day 1 | -1.06 (0.625) | -0.23 (0.486)
  Change from Predose at 360 min Postdose on Day 1: number analyzed (Participants) | 39 | 20
  Change from Predose at 360 min Postdose on Day 1 | -0.78 (0.517) | -0.10 (0.440)
  Change from Predose at 480 min Postdose on Day 1: number analyzed (Participants) | 39 | 19
  Change from Predose at 480 min Postdose on Day 1 | -0.63 (0.570) | -0.13 (0.459)
  Predose on Day 15: number analyzed (Participants) | 37 | 20
  Predose on Day 15 | 1.57 (0.645) | 1.24 (0.349)
  Change from Predose at 1 min Postdose on Day 15: number analyzed (Participants) | 37 | 19
  Change from Predose at 1 min Postdose on Day 15 | -0.78 (0.496) | -0.16 (0.279)
  Change from Predose at 5 min Postdose on Day 15: number analyzed (Participants) | 37 | 19
  Change from Predose at 5 min Postdose on Day 15 | -1.03 (0.569) | -0.25 (0.354)
  Predose on Day 29: number analyzed (Participants) | 36 | 19
  Predose on Day 29 | 1.64 (0.461) | 1.36 (0.304)
  Change from Predose at 1 min Postdose on Day 29: number analyzed (Participants) | 36 | 19
  Change from Predose at 1 min Postdose on Day 29 | -0.88 (0.469) | -0.24 (0.306)
  Change from Predose at 5 min Postdose on Day 29: number analyzed (Participants) | 36 | 19
  Change from Predose at 5 min Postdose on Day 29 | -1.21 (0.416) | -0.37 (0.347)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 36
Description: All randomized participants who received at least 1 dose of study drug (Safety Population).
Arm/Group | Brimonidine Tartrate | Brimonidine Tartrate Vehicle
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 10/40 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brimonidine Tartrate (N=40) | Brimonidine Tartrate Vehicle (N=20)
Bronchitis (Infections and infestations) | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.